CLINICAL TRIAL: NCT04956575
Title: A Phase 1/2, Randomized, Stratified, Observer-Blind, Dose-Ranging Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1010 Seasonal Influenza Vaccine in Healthy Adults 18 Years and Older
Brief Title: A Study of mRNA-1010 Seasonal Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1010-P101
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Seasonal Influenza
Keywords: Influenza vaccine; mRNA-1010; Moderna
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1010 influenza vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Phase 1/2: mRNA-1010 Dose Level A (Experimental): Participants will receive mRNA-1010 at dose level A by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 1/2: mRNA-1010 Dose Level B (Experimental): Participants will receive mRNA-1010 at dose level B by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 1/2: mRNA-1010 Dose Level C (Experimental): Participants will receive mRNA-1010 at dose level C by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 1/2: Placebo (Experimental): Participants will receive placebo matching to mRNA-1010 by IM injection on Day 1.
  Interventions: Biological: Placebo
- Phase 2 NH: Active Comparator Dose Level A (Active Comparator): Participants will receive active comparator at dose level A by IM injection on Day 1.
  Interventions: Biological: Active Comparator
- Phase 2 NH: mRNA-1010 Dose Level D (Experimental): Participants will receive mRNA-1010 at dose level D by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 2 NH: mRNA-1010 Dose Level A (Experimental): Participants will receive mRNA-1010 at dose level A by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 2 NH: mRNA-1010 Dose Level B (Experimental): Participants will receive mRNA-1010 at dose level B by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 2 Extension: Active Comparator Dose Level A (Active Comparator): Participants will receive active comparator at dose level A by IM injection on Day 1.
  Interventions: Biological: Active Comparator
- Phase 2 Extension: mRNA-1010 Dose Level D (Experimental): Participants will receive mRNA-1010 at dose level D by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 2 Extension: mRNA-1010 Dose Level E (Experimental): Participants will receive mRNA-1010 at dose level E by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- Phase 2 Extension: mRNA-1010 Dose Level F (Experimental): Participants will receive mRNA-1010 at dose level F by IM injection on Day 1.
  Interventions: Biological: mRNA-1010

INTERVENTIONS:
Biological: mRNA-1010 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: Phase 1/2: mRNA-1010 Dose Level A; Phase 1/2: mRNA-1010 Dose Level B; Phase 1/2: mRNA-1010 Dose Level C; Phase 2 Extension: mRNA-1010 Dose Level D; Phase 2 Extension: mRNA-1010 Dose Level E; Phase 2 Extension: mRNA-1010 Dose Level F; Phase 2 NH: mRNA-1010 Dose Level A; Phase 2 NH: mRNA-1010 Dose Level B; Phase 2 NH: mRNA-1010 Dose Level D
Biological: Placebo — 0.9% sodium chloride solution for injection
  Arms: Phase 1/2: Placebo
Biological: Active Comparator — 0.5 milliliter (mL) intramuscular (IM) injection
  Other Names: Licensed quadrivalent seasonal influenza
  Arms: Phase 2 Extension: Active Comparator Dose Level A; Phase 2 NH: Active Comparator Dose Level A

SUMMARY:
The study comprises 3 parts: Phase 1/2, Phase 2 Northern Hemisphere (NH), and Phase 2 extension. The primary objective of this study is to evaluate the safety, reactogenicity, and humoral immunogenicity of mRNA-1010 vaccine.

ELIGIBILITY:
Key Inclusion Criteria:

Phase 1/2:

* Participant has a body mass index (BMI) of 18 kilograms (kg)/square meter (m^2) to 35 kg/m^2 (inclusive) at the Screening Visit.
* Participant is in good health, in the opinion of the Investigator, based on review of medical history and physical examination performed at screening.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 3 months following vaccine administration, and not currently breastfeeding.

Phase 2 NH and Phase 2 Extension:

* Participant is medically stable, in the opinion of the Investigator, based on review of medical history and physical examination performed at screening.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 3 months following vaccine administration, and not currently breastfeeding.

Key Exclusion Criteria:

Phase 1/2:

* Participant has had significant exposure to someone with laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, COVID-19, or influenza-like illness (ILI) in the past 14 days prior to the Screening Visit, as defined by the United States Centers for Disease Control and Prevention (CDC) as close contact with someone who has COVID-19.
* Participant has a positive SARS-CoV-2 reverse transcriptase polymerase chain reaction (RT-PCR) or antigen test in the past 10 days prior to the Screening Visit.
* Participant is acutely ill or febrile (body temperature ≥ 38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Participant has a pre-existing medical condition that is not stable, at the discretion of the Investigator.
* Participant has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment.
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening Visit (for corticosteroids ≥10 milligrams [mg]/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Participant has received or plans to receive any licensed vaccine ≤28 days prior to the investigational product (IP) injection (Day 1) or plans to receive a licensed vaccine within 28 days after the IP injection, with the exception of vaccines authorized or approved for the prevention of COVID-19 (regardless of type of vaccine) that become available to participants during the study. Efforts should be made to space study vaccination and COVID-19 vaccination by at least 7 and preferably 14 days, but COVID-19 vaccination should not be delayed.
* Participant has received a seasonal influenza vaccine or any other investigational influenza vaccine after 01 January 2021.

Phase 2 NH:

* Participant has had close contact to someone with SARS-CoV-2 infection or COVID-19 as defined by the CDC (CDC 2021a) in the past 14 days prior to the Screening Visit, unless the participant has been fully vaccinated for COVID-19.
* Participant is acutely ill or febrile (body temperature ≥ 38.0°C/100.4°F) 72 hours prior to or at the Screening Visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day screening window and will retain their initially assigned participant number.
* Participant has a medical, psychiatric, occupational condition, or history of substance abuse that may pose additional risk as a result of participation or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment.
* Participant has a current or previous diagnosis of immunocompromising/immunosuppressive condition, immune mediated disease requiring immune-modifying therapy, asplenia, recurrent severe infections (human immunodeficiency virus [HIV] positive participants on antiretroviral therapy with cluster of differentiation [CD] 4 count ≥ 350 cells/mm3 and HIV RNA ≤ 500 copies/mL within the past 12 months are permitted).
* Participant has received systemic immunosuppressants or immune-modifying drugs for > 14 days in total within 6 months prior to Screening Visit (for corticosteroids ≥ 10 mg/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study.
* Participant has a history of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine or any of the components contained in the mRNA 1010 or the comparator vaccine, which is an egg-based influenza vaccine.
* Participant has received or plans to receive any licensed vaccine ≤ 28 days prior to the IP injection (Day 1) or plans to receive a licensed vaccine within 28 days after the IP injection, with the exception of vaccines authorized or approved for the prevention of COVID-19 (regardless of type of vaccine) that become available to participants during the study. Efforts should be made to space study vaccination and COVID-19 vaccination by at least 7 and preferably 14 days, but COVID-19 vaccination should not be delayed.
* Participant has received a seasonal influenza vaccine or any other investigational influenza vaccine within 6 months prior to the Screening Visit.
* Participant has tested positive for influenza by CDC-recommended testing methods within 6 months prior to the Screening Visit.
* Participant has participated in an interventional clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.

Phase 2 Extension:

* Participant has had close contact to someone with SARS-CoV-2 infection or COVID-19 as defined by the CDC in the past 10 days prior to the Screening Visit.
* Participant is acutely ill or febrile (body temperature ≥ 38.0°C/100.4°F) 72 hours prior to or at the Screening Visit or Day 1. Participants meeting this criterion may be rescheduled within the 28-day screening window and will retain their initially assigned participant number.
* Participant has a medical, psychiatric, occupational condition, or history of substance abuse that may pose additional risk as a result of participation or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment.
* Participant has a current or previous diagnosis of immunocompromising/immunosuppressive condition, immune-mediated disease requiring immune-modifying therapy, asplenia, recurrent severe infections (HIV-positive participants on antiretroviral therapy with CD 4 count ≥ 350 cells/mm^3 and HIV-RNA ≤ 500 copies/mL within the past 365 days are permitted).
* Participant has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 180 days prior to Screening Visit (for corticosteroids ≥ 10 mg/day of prednisone or equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study.
* Participant has a history of anaphylaxis, urticaria, or other significant AR requiring medical intervention after receipt of a vaccine or any of the components contained in the mRNA-1010 or the comparator vaccine, which is an egg-based influenza vaccine.
* Participant has received or plans to receive any licensed vaccine ≤ 28 days prior to the IP injection (Day 1) or plans to receive a licensed vaccine within 28 days after the IP injection, with the exception of vaccines authorized or approved for the prevention of COVID-19 (regardless of type of vaccine) that become available to participants during the study. Efforts should be made to space study vaccination and COVID-19 vaccination by at least 7 and preferably 14 days, but COVID-19 vaccination should not be delayed.
* Participant has received a seasonal influenza vaccine or any other investigational influenza vaccine within 180 days prior to the randomization visit.
* Participant had tested positive for influenza by CDC-recommended testing methods within 180 days prior to the Screening Visit.
* Participant has participated in an interventional clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Cognitive Clinical Trials - Phoenix, Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC - Phoenix, Tempe, Arizona
  - Benchmark Research - Colton, CA, Colton, California
  - Research Centers of America - ERGG - PPDS, Hollywood, Florida
  - Meridian Clinical Research (Savannah Georgia) - Platinum - PPDS, Savannah, Georgia
  - Meridian Clinical Research, Sioux City, Iowa
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Meridian Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - Meridian Clinical Research, Rockville, Maryland
  - Meridian Clinical Research (Grand Island), Grand Island, Nebraska
  - Meridian Clinical Research, LLC (Lincoln Nebraska), Lincoln, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research (Endwell-New York) - Platinum - PPDS, Endwell, New York
  - Lucas Research, Morehead City, North Carolina
  - Trial Management Associates LLC - ERN - PPDS, Wilmington, North Carolina
  - Meridian Clinical Research - Cincinnati - Platinum - PPDS, Cincinnati, Ohio
  - Keystone VitaLink Research - Greenville - PPDS, Greenville, South Carolina
  - PanAmerican Clinical Research LLC, Brownsville, Texas
  - Research Your Health - ERN - PPDS, Plano, Texas
  - South Ogden Family Medicine/Ogden Clinic - CCT, South Ogden, Utah

REFERENCES:
- [Result] Lee IT, Nachbagauer R, Ensz D, Schwartz H, Carmona L, Schaefers K, Avanesov A, Stadlbauer D, Henry C, Chen R, Huang W, Schrempp DR, Ananworanich J, Paris R. Safety and immunogenicity of a phase 1/2 randomized clinical trial of a quadrivalent, mRNA-based seasonal influenza vaccine (mRNA-1010) in healthy adults: interim analysis. Nat Commun. 2023 Jun 19;14(1):3631. doi: 10.1038/s41467-023-39376-7. PMID 37336877
- [Derived] Ananworanich J, Lee IT, Ensz D, Carmona L, Schaefers K, Avanesov A, Stadlbauer D, Choi A, Pucci A, McGrath S, Kuo HH, Henry C, Chen R, Huang W, Nachbagauer R, Paris R. Safety and Immunogenicity of mRNA-1010, an Investigational Seasonal Influenza Vaccine, in Healthy Adults: Final Results From a Phase 1/2 Randomized Trial. J Infect Dis. 2025 Feb 4;231(1):e113-e122. doi: 10.1093/infdis/jiae329. PMID 38934845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 20 centers in the United States. The vaccines used in the study were based on the influenza virus strains recommended by the World Health Organization for the southern and northern hemispheres.
Pre-assignment Details: For Phase 1/2, 1 participant who was randomly assigned to the 200 micrograms (ug) mRNA-1010 group received a dose of 100 ug and was therefore included in the 100 ug mRNA-1010 group in the Safety Set and the Solicited Safety Set.
  For Phase 2 Northern Hemisphere (NH), 1 participant randomly assigned to the 25 ug mRNA-1010 group received 50 ug mRNA-1010, and 1 participant randomly assigned to 50 ug mRNA-1010 received Afluria Quadrivalent.
Groups:
- Phase 1/2: Placebo: Participants received placebo matching to mRNA-1010 by intramuscular (IM) injection on Day 1.
- Phase 1/2: mRNA-1010 50 ug; Phase 2 NH: mRNA-1010 50 ug: Participants received mRNA-1010 50 ug by IM injection on Day 1.
- Phase 1/2: mRNA-1010 100 ug; Phase 2 NH: mRNA-1010 100 ug: Participants received mRNA-1010 100 ug by IM injection on Day 1.
- Phase 1/2: mRNA-1010 200 ug: Participants received mRNA-1010 200 ug by IM injection on Day 1.
- Phase 2 NH: Afluria Quadrivalent 60 ug; Phase 2 Extension: Afluria Quadrivalent 60 ug: Participants received Afluria Quadrivalent 60 ug by IM injection on Day 1.
- Phase 2 NH: mRNA-1010 25 ug; Phase 2 Extension: mRNA-1010 25 ug: Participants received mRNA-1010 25 ug by IM injection on Day 1.
- Phase 2 Extension: mRNA-1010 6.25 ug: Participants received mRNA-1010 6.25 ug by IM injection on Day 1.
- Phase 2 Extension: mRNA-1010 12.5 ug: Participants received mRNA-1010 12.5 ug by IM injection on Day 1.
Period: Overall Study
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug | Phase 2 Extension: Afluria Quadrivalent 60 ug | Phase 2 Extension: mRNA-1010 6.25 ug | Phase 2 Extension: mRNA-1010 12.5 ug | Phase 2 Extension: mRNA-1010 25 ug
Started | 45 | 45 | 45 | 45 | 53 | 153 | 149 | 148 | 51 | 50 | 51 | 50
Received at Least 1 Dose of Investigational Product (Numbers are based on planned vaccination group.) | 45 | 45 | 45 | 45 | 53 | 151 | 147 | 147 | 51 | 50 | 50 | 49
Safety Analysis Set (Safety Analysis Set consisted of all randomly assigned participants who received the investigational product. The Safety Set was used for analysis of safety except for the solicited adverse reactions (ARs). Participants were included in the vaccination group corresponding to the study injection they actually received.) | 45 | 45 | 46 | 44 | 54 | 150 | 147 | 147 | 51 | 50 | 50 | 49
Solicited Safety Set (Solicited Safety Set consisted of all participants in the Safety Set who contributed any solicited AR data. Participants were included in the vaccination group corresponding to the study injection they actually received.) | 44 | 45 | 46 | 44 | 53 | 149 | 146 | 145 | 51 | 50 | 50 | 49
Per-Protocol (PP) Set (PP Set consisted of all participants who received the investigational product and who complied with the injection schedule and timing of immunogenicity blood sampling, did not have influenza infection at baseline through Day 29, and had no major protocol deviations that impacted the immune response.) | 41 | 43 | 44 | 41 | 52 | 144 | 138 | 141 | 48 | 49 | 47 | 46
Completed (Participants were considered to have completed the study if they completed the final visit on Day 181 (Month 6), 6 months after the investigational product administration on Day 1) | 40 | 39 | 42 | 38 | 50 | 135 | 133 | 139 | 46 | 47 | 45 | 41
Not Completed | 5 | 6 | 3 | 7 | 3 | 18 | 16 | 9 | 5 | 3 | 6 | 9
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 2 | 3 | 1 | 10 | 11 | 7 | 4 | 2 | 3 | 8
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 4 | 2 | 8 | 5 | 1 | 1 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: All randomly assigned participants who received the investigational product.
Groups:
- Phase 1/2: Placebo: Participants received placebo matching to mRNA-1010 by IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug | Phase 2 Extension: Afluria Quadrivalent 60 ug | Phase 2 Extension: mRNA-1010 6.25 ug | Phase 2 Extension: mRNA-1010 12.5 ug | Phase 2 Extension: mRNA-1010 25 ug | Total
Number analyzed (Participants) | 45 | 45 | 46 | 44 | 54 | 150 | 147 | 147 | 51 | 50 | 50 | 49 | 878
Age, Continuous [Mean (Full Range); unit: years] | 52.0 [18 to 90] | 48.2 [18 to 74] | 52.2 [19 to 83] | 48.9 [19 to 89] | 52.4 [20 to 86] | 50.4 [18 to 86] | 50.3 [19 to 81] | 49.9 [18 to 82] | 40.8 [19 to 65] | 40.4 [18 to 75] | 42.8 [19 to 76] | 38.9 [21 to 74] | 47.3 [18 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 25 | 33 | 30 | 89 | 80 | 86 | 24 | 34 | 27 | 30 | 500
  Male | 22 | 26 | 21 | 11 | 24 | 61 | 67 | 61 | 27 | 16 | 23 | 19 | 378
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 9 | 8 | 12 | 27 | 32 | 29 | 17 | 12 | 14 | 11 | 188
  Not Hispanic or Latino | 39 | 33 | 37 | 35 | 42 | 122 | 114 | 114 | 34 | 36 | 35 | 36 | 677
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 2 | 1 | 2 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38 | 38 | 41 | 32 | 45 | 124 | 120 | 124 | 47 | 44 | 39 | 41 | 733
  Black or African American | 5 | 5 | 2 | 10 | 6 | 17 | 18 | 18 | 4 | 4 | 8 | 4 | 101
  Asian | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 2 | 0 | 12
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Multiple Race | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 1 | 0 | 1 | 1 | 1 | 11
  Other Race | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 4
  Race Not Reported | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 10
  Race Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic ARs
Description: Solicited ARs (local and systemic) were collected in the electronic diary (eDiary). Local ARs included: pain at injection site, erythema (redness) at injection site, swelling/induration (hardness) at injection site, and localized axillary swelling or tenderness ipsilateral to the injection arm. Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, rash, body temperature (potentially fever), and chills. Solicited ARs (local and systemic) considered causally related to injection were graded 0-4; lower score indicates lower severity and a higher score indicates greater severity. Note, not all solicited ARs were considered adverse events (AEs). The Investigator reviewed whether the solicited AR was also to be recorded as an AE. Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is in Reported "Adverse Events" section and presented by Phase/dose group.
Time Frame: 7 days after vaccination
Population: Solicited Safety Set: Consisted of all participants in the Safety Set who contributed any solicited AR data. Dose groups for Phase 1/2, Phase 2 NH, and Phase 2 Extension by dose group and Afluria Quadrivalent 60 ug groups were combined for this assessment as pre-specified by the protocol. Combined data for >= 50 ug is also presented. Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received placebo matching to mRNA-1010 by IM injection on Day 1.
- Afluria Quadrivalent 60 ug: Participants received Afluria Quadrivalent 60 ug by IM injection on Day 1.
- mRNA-1010 6.25 ug: Participants received mRNA-1010 6.25 ug by IM injection on Day 1.
- mRNA-1010 12.5 ug: Participants received mRNA-1010 12.5 ug by IM injection on Day 1.
- mRNA-1010 25 ug: Participants received mRNA-1010 25 ug by IM injection on Day 1.
- mRNA-1010 50 ug: Participants received mRNA-1010 50 ug by IM injection on Day 1.
- mRNA-1010 100 ug: Participants received mRNA-1010 100 ug by IM injection on Day 1.
- mRNA-1010 200 ug: Participants received mRNA-1010 200 ug by IM injection on Day 1.
- mRNA-1010 >= 50 ug Overall: Participants received mRNA-1010 >= 50 ug by IM injection on Day 1.
Arm/Group | Placebo | Afluria Quadrivalent 60 ug | mRNA-1010 6.25 ug | mRNA-1010 12.5 ug | mRNA-1010 25 ug | mRNA-1010 50 ug | mRNA-1010 100 ug | mRNA-1010 200 ug | mRNA-1010 >= 50 ug Overall
Number analyzed (Participants) | 44 | 104 | 50 | 50 | 198 | 191 | 191 | 44 | 426
Participants
  Grade 1 | 12 | 43 | 22 | 16 | 76 | 65 | 44 | 7 | 116
  Grade 2 | 5 | 16 | 17 | 12 | 81 | 70 | 86 | 17 | 173
  Grade 3 | 1 | 4 | 4 | 4 | 15 | 31 | 45 | 18 | 94
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. A treatment-emergent AE (TEAE) was defined as any event not present before exposure to vaccine or any event already present that worsens in intensity or frequency after exposure. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsens from baseline and is considered clinically significant in the medical and scientific judgment of the Investigator. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study, regardless of causality, is located in the Reported "Adverse Events" section and presented by each Phase and dose group separately.
Time Frame: Up to 28 days after vaccination
Population: Safety Analysis Set: all randomly assigned participants who received the investigational product. Dose groups for Phase 1/2, Phase 2 NH, and Phase 2 Extension by dose group and Afluria Quadrivalent 60 ug groups were combined for this assessment as pre-specified by the protocol. Combined data for >= 50 ug is also presented. Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Afluria Quadrivalent 60 ug | mRNA-1010 6.25 ug | mRNA-1010 12.5 ug | mRNA-1010 25 ug | mRNA-1010 50 ug | mRNA-1010 100 ug | mRNA-1010 200 ug | mRNA-1010 >= 50 ug Overall
Number analyzed (Participants) | 45 | 105 | 50 | 50 | 199 | 192 | 193 | 44 | 429
Participants
  All | 6 | 20 | 17 | 14 | 47 | 42 | 46 | 10 | 98
  Serious | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 3
  Nonserious | 5 | 20 | 16 | 14 | 47 | 41 | 44 | 10 | 95

3. Primary Outcome: Number of Participants With SAEs, AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs)
Description: An SAE was defined as any AE that resulted in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event.
  AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis.
  An MAAE is an AE that leads to an unscheduled visit to an healthcare practitioner. This would include visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or COVID-19 and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section and presented by each Phase and dose group separately.
Time Frame: Up to 6 months (end of study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- mRNA-1010 25 ug: Participants receive mRNA-1010 25 ug by IM injection on Day 1.
- mRNA-1010 50 ug: Participants receive mRNA-1010 50 ug by IM injection on Day 1.
- mRNA-1010 >= 50 ug: Participants received mRNA-1010 mRNA-1010 >= 50 ug by IM injection on Day 1.
Arm/Group | Placebo | Afluria Quadrivalent 60 ug | mRNA-1010 6.25 ug | mRNA-1010 12.5 ug | mRNA-1010 25 ug | mRNA-1010 50 ug | mRNA-1010 100 ug | mRNA-1010 200 ug | mRNA-1010 >= 50 ug
Number analyzed (Participants) | 45 | 105 | 50 | 50 | 199 | 192 | 193 | 44 | 429
Participants
  SAE | 2 | 2 | 2 | 0 | 3 | 5 | 4 | 1 | 10
  AESI | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MAAE | 10 | 27 | 18 | 15 | 58 | 50 | 62 | 12 | 124

4. Primary Outcome: Phase 1/2: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies at Day 29, as Measured by Hemagglutination Inhibition (HAI) Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. GMT 95% confidence interval (CI) was calculated based on the t-distribution of the log-transformed values then back transformed to the original scale for presentation.
Time Frame: Day 29
Population: Per-Protocol (PP) Set: consisted of all participants who received the investigational product and who complied with the injection schedule and timing of immunogenicity blood sampling, did not have influenza infection at baseline through Day 29, and had no major protocol deviations that impacted the immune response. Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug
Number analyzed (Participants) | 41 | 43 | 44 | 41
Titer
  H1N1 | 58.50 [39.17 to 87.38] | 410.71 [262.55 to 642.47] | 331.06 [214.34 to 511.34] | 598.22 [370.14 to 966.84]
  H3N2 | 56.49 [38.27 to 83.36] | 376.02 [272.52 to 518.81] | 325.07 [234.58 to 450.47] | 537.26 [386.28 to 747.26]
  Victoria-lineage | 111.14 [75.41 to 163.80] | 237.44 [178.78 to 315.34] | 169.92 [122.03 to 236.60] | 281.00 [213.37 to 370.06]
  Yamagata-lineage | 103.94 [66.83 to 161.65] | 379.02 [277.02 to 518.57] | 319.07 [218.60 to 465.73] | 456.36 [341.14 to 610.50]

5. Primary Outcome: Phase 2 NH: GMT of HA Antibodies at Day 29, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: Humoral immunogenicity relative to that of the active comparator (afluria quadrivalent) was assessed against vaccine-matched Influenza A and B strains at Day 29. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. GMT 95% CI was calculated based on the t-distribution of the log-transformed values then back transformed to the original scale for presentation.
Time Frame: Day 29
Population: PP Set: consisted of all participants who received the investigational product and who complied with the injection schedule and timing of immunogenicity blood sampling, did not have influenza infection at baseline through Day 29, and had no major protocol deviations that impacted the immune response. Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug
Number analyzed (Participants) | 52 | 144 | 138 | 141
titer
  H1N1 | 164.00 [120.18 to 223.81] | 298.88 [247.21 to 361.36] | 422.24 [347.72 to 512.73] | 443.62 [366.58 to 536.85]
  H3N2 | 85.54 [64.33 to 113.74] | 153.43 [128.99 to 182.50] | 187.08 [156.64 to 223.43] | 215.23 [180.75 to 256.28]
  Victoria-lineage | 147.47 [119.98 to 181.24] | 100.51 [88.63 to 114.00] | 129.56 [113.92 to 147.36] | 123.17 [108.47 to 139.85]
  Yamagata-lineage | 193.08 [155.16 to 240.27] | 215.19 [188.30 to 245.92] | 230.66 [201.23 to 264.40] | 231.44 [202.38 to 264.68]
Statistical Analysis 1: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.82, 95% CI 2-sided [1.27 to 2.61] — The 2 sided 95% assessed the difference in immune response between the mRNA-1010 compared with the active comparator, Afluria Quadrivalent, at Day 29
Statistical Analysis 2: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 2.57, 95% CI 2-sided [1.79 to 3.70] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 2.70, 95% CI 2-sided [1.88 to 3.88] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.79, 95% CI 2-sided [1.29 to 2.50] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 2.19, 95% CI 2-sided [1.57 to 3.05] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 2.52, 95% CI 2-sided [1.81 to 3.50] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.68, 95% CI 2-sided [0.54 to 0.87] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.88, 95% CI 2-sided [0.69 to 1.12] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.84, 95% CI 2-sided [0.66 to 1.06] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.11, 95% CI 2-sided [0.86 to 1.44] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.19, 95% CI 2-sided [0.93 to 1.54] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.20, 95% CI 2-sided [0.93 to 1.55] — [estimate comment as in outcome 5, analysis 1]

6. Primary Outcome: Phase 2 Extension: GMT of HA Antibodies at Day 29, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: as for outcome 5
Time Frame: Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Phase 2 Extension: Afluria Quadrivalent 60 ug | Phase 2 Extension: mRNA-1010 6.25 ug | Phase 2 Extension: mRNA-1010 12.5 ug | Phase 2 Extension: mRNA-1010 25 ug
Number analyzed (Participants) | 48 | 49 | 47 | 46
Titer
  H1N1 | 253.07 [180.86 to 354.12] | 228.02 [163.17 to 318.64] | 316.53 [225.12 to 445.06] | 471.56 [334.39 to 664.99]
  H3N2 | 114.21 [82.80 to 157.55] | 161.58 [117.46 to 222.27] | 216.32 [156.34 to 299.30] | 301.53 [217.28 to 418.45]
  Victoria-lineage: number analyzed (Participants) | 48 | 49 | 46 | 46
  Victoria-lineage | 155.07 [121.65 to 197.66] | 55.76 [43.81 to 70.97] | 71.12 [55.51 to 91.11] | 83.46 [65.16 to 106.90]
  Yamagata-lineage: number analyzed (Participants) | 48 | 49 | 46 | 46
  Yamagata-lineage | 193.16 [147.41 to 253.12] | 119.54 [91.34 to 156.45] | 178.43 [135.33 to 235.26] | 144.13 [109.16 to 190.29]
Statistical Analysis 1: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.90, 95% CI 2-sided [0.57 to 1.44] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.25, 95% CI 2-sided [0.78 to 2.00] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent. against H1N1 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.86, 95% CI 2-sided [1.16 to 2.99] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.41, 95% CI 2-sided [0.91 to 2.21] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 1.89, 95% CI 2-sided [1.21 to 2.97] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 2.64, 95% CI 2-sided [1.68 to 4.14] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.36, 95% CI 2-sided [0.26 to 0.50] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.46, 95% CI 2-sided [0.33 to 0.64] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.54, 95% CI 2-sided [0.38 to 0.76] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.62, 95% CI 2-sided [0.43 to 0.90] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.92, 95% CI 2-sided [0.63 to 1.35] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: Phase 2 Extension: Afluria Quadrivalent 60 ug vs Phase 2 Extension: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other — The ratio of GMT was estimated by the ratio of model based GMT; Ratio = 0.75, 95% CI 2-sided [0.51 to 1.09] — [estimate comment as in outcome 5, analysis 1]

7. Primary Outcome: Phase 1/2: Percentage of Participants With Seroconversion, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B
Description: Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
  Seroconversion at a participant level was defined as (a) if lower limit of quantification (LLOQ) was 1:10, a post-baseline titer ≥1:40 if baseline was <1:10 or a 4-fold or greater rise from baseline if baseline was ≥1:10 in anti-HA antibodies; or (b) if LLOQ was >1:10, a post-baseline titer ≥4 x LLOQ if baseline was <LLOQ, or 4-fold or greater increase from baseline if baseline was ≥LLOQ in anti-HA antibodies.
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug
Number analyzed (Participants) | 41 | 43 | 44 | 41
percentage of participants
  H1N1 | 4.9 [0.60 to 16.53] | 67.4 [51.46 to 80.92] | 81.8 [67.29 to 91.81] | 90.2 [76.87 to 97.28]
  H3N2 | 2.4 [0.06 to 12.86] | 81.4 [66.60 to 91.61] | 75.0 [59.66 to 86.81] | 75.6 [59.70 to 87.64]
  Victoria-lineage: number analyzed (Participants) | 41 | 43 | 44 | 40
  Victoria-lineage | 2.4 [0.06 to 12.86] | 14.0 [5.30 to 27.93] | 15.9 [6.64 to 30.07] | 25.0 [12.69 to 41.20]
  Yamagata-lineage | 2.4 [0.06 to 12.86] | 41.9 [27.01 to 57.87] | 50.0 [34.56 to 65.44] | 51.2 [35.13 to 67.12]

8. Primary Outcome: Phase 1/2: Geometric Mean Fold-Rise (GMFR) of Anti-HA Antibodies at Day 29, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
  95% CI was calculated based on the difference in the log-transformed values for GMFR, then back transformed to the original scale for presentation.
Time Frame: Day 1 (Baseline), Day 29
Population: PP Set: consisted of all participants who received the investigational product and who complied with the injection schedule and timing of immunogenicity blood sampling, did not have influenza infection at baseline through Day 29, and had no major protocol deviations that impacted the immune response.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug
Number analyzed (Participants) | 41 | 43 | 44 | 41
ratio
  H1N1 | 1.08 [0.91 to 1.29] | 7.50 [5.00 to 11.26] | 8.69 [6.03 to 12.50] | 11.05 [7.59 to 16.11]
  H3N2 | 1.05 [0.80 to 1.39] | 7.16 [5.19 to 9.88] | 6.43 [4.54 to 9.10] | 7.13 [5.12 to 9.93]
  Victoria-lineage | 0.98 [0.80 to 1.20] | 1.95 [1.61 to 2.37] | 1.86 [1.36 to 2.53] | 2.03 [1.50 to 2.75]
  Yamagata-lineage | 0.92 [0.81 to 1.05] | 3.04 [2.34 to 3.96] | 3.78 [2.70 to 5.28] | 3.55 [2.47 to 5.11]

9. Primary Outcome: Phase 2 NH: Percentage of Participants With Seroconversion, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B
Description: Humoral immunogenicity relative to that of the active comparator (afluria quadrivalent) was assessed against vaccine-matched Influenza A and B strains at Day 29. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
  Seroconversion at a participant level was defined as (a) if LLOQ was 1:10, a post-baseline titer ≥1:40 if baseline was <1:10 or a 4-fold or greater rise from baseline if baseline was ≥1:10 in anti-HA antibodies; or (b) if LLOQ was >1:10, a post-baseline titer ≥4 x LLOQ if baseline was <LLOQ, or 4-fold or greater increase from baseline if baseline was ≥LLOQ in anti-HA antibodies.
  95% CI was calculated using the Clopper-Pearson method
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug
Number analyzed (Participants) | 52 | 144 | 138 | 141
percentage of participants
  H1N1 | 59.6 [45.10 to 72.99] | 72.2 [64.15 to 79.36] | 84.8 [77.68 to 90.33] | 85.8 [78.95 to 91.12]
  H3N2 | 40.4 [27.01 to 54.90] | 66.0 [57.62 to 73.65] | 71.7 [63.45 to 79.07] | 78.7 [71.04 to 85.16]
  Victoria-lineage: number analyzed (Participants) | 52 | 144 | 138 | 140
  Victoria-lineage | 32.7 [20.33 to 47.11] | 22.9 [16.33 to 30.65] | 33.3 [25.54 to 41.86] | 37.1 [29.13 to 45.71]
  Yamagata-lineage | 32.7 [20.33 to 47.11] | 41.7 [33.52 to 50.17] | 47.8 [39.26 to 56.49] | 51.8 [43.21 to 60.26]
Statistical Analysis 1: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other; Percent difference = 12.61, 95% CI 2-sided [-2.00 to 27.93] — Seroconversion percent difference of mRNA-1010 - Afluria Quadrivalent. 95% CI was calculated using the Miettinen-Nurminen (score) method
Statistical Analysis 2: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other; Percent difference = 25.17, 95% CI 2-sided [11.18 to 39.89] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other; Percent Difference = 26.20, 95% CI 2-sided [12.33 to 40.84] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other; Percent Difference = 25.59, 95% CI 2-sided [9.82 to 40.13] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other; Percent Difference = 31.35, 95% CI 2-sided [15.66 to 45.73] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other; Percent Difference = 38.34, 95% CI 2-sided [22.98 to 52.30] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other; Percent Difference = -9.78, 95% CI 2-sided [-24.83 to 3.79] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other; Percent Difference = 0.64, 95% CI 2-sided [-14.91 to 14.73] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other; Percent Difference = 4.45, 95% CI 2-sided [-11.19 to 18.59] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other; Percent Difference = 8.97, 95% CI 2-sided [-6.72 to 23.09] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 50 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other; Percent Difference = 15.13, 95% CI 2-sided [-0.74 to 29.37] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: Phase 2 NH: Afluria Quadrivalent 60 ug vs Phase 2 NH: mRNA-1010 100 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent. against Yamagata-lineage at Day 29; Test type: Other; Percent Difference = 19.08, 95% CI 2-sided [3.22 to 33.22] — [estimate comment as in outcome 9, analysis 1]

10. Primary Outcome: Phase 2 Extension: Percentage of Participants With Seroconversion, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B
Description: as for outcome 9
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Afluria Quadrivalent 60 ug | mRNA-1010 6.25 ug | mRNA-1010 12.5 ug | mRNA-1010 25 ug
Number analyzed (Participants) | 48 | 49 | 47 | 46
percentage of participants
  H1N1 | 50.0 [35.23 to 64.77] | 59.2 [44.21 to 73.00] | 68.1 [52.88 to 80.91] | 73.9 [58.87 to 85.73]
  H3N2 | 43.8 [29.48 to 58.82] | 44.9 [30.67 to 59.77] | 66.0 [50.69 to 79.14] | 80.4 [66.09 to 90.64]
  Victoria-lineage | 47.9 [33.29 to 62.81] | 10.2 [3.40 to 22.23] | 21.7 [10.95 to 36.36] | 28.3 [15.99 to 43.46]
  Yamagata-lineage | 47.9 [33.29 to 62.81] | 24.5 [13.34 to 38.87] | 43.5 [28.93 to 58.89] | 39.1 [25.09 to 54.63]
Statistical Analysis 1: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other; Percent Difference = 9.18, 95% CI 2-sided [-10.62 to 28.31] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other; Percent Difference = 18.09, 95% CI 2-sided [-1.81 to 36.61] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H1N1 at Day 29; Test type: Other; Percent Difference = 23.91, 95% CI 2-sided [4.20 to 41.86] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other; Percent Difference = 1.15, 95% CI 2-sided [-18.41 to 20.60] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other; Percent Difference = 22.21, 95% CI 2-sided [2.09 to 40.60] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against H3N2 at Day 29; Test type: Other; Percent Difference = 36.68, 95% CI 2-sided [17.38 to 53.36] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other; Percent Difference = -37.71, 95% CI 2-sided [-53.36 to -20.45] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other; Treatment Difference = -26.18, 95% CI 2-sided [-43.66 to -6.90] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Victoria-lineage at Day 29; Test type: Other; Percent Difference = -19.66, 95% CI 2-sided [-37.95 to 0.11] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 6.25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other; Percent Difference = -23.43, 95% CI 2-sided [-41.09 to -4.26] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 12.5 ug; Humoral immunogenicity of mRNA-1010 relative to that of against Afluria Quadrivalent Yamagata-lineage at Day 29; Test type: Other; Percent Difference = -4.44, 95% CI 2-sided [-24.09 to 15.59] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: Afluria Quadrivalent 60 ug vs mRNA-1010 25 ug; Humoral immunogenicity of mRNA-1010 relative to that of Afluria Quadrivalent against Yamagata-lineage at Day 29; Test type: Other; Percent Difference = -8.79, 95% CI 2-sided [-28.13 to 11.27] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Phase 1/2: GMT of Anti-HA Antibodies at Days 1, 8 and 181, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. GMT 95% CI was calculated based on the t-distribution of the log-transformed values then back transformed to the original scale for presentation.
Time Frame: Day 1 (Baseline), Day 8 and Day 181
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug
Number analyzed (Participants) | 41 | 43 | 44 | 41
titer
  Day 1 (Baseline): H1N1 | 54.16 [35.85 to 81.83] | 54.73 [37.76 to 79.31] | 38.12 [28.35 to 51.26] | 54.12 [37.26 to 78.61]
  Day 8: H1N1: number analyzed (Participants) | 41 | 42 | 44 | 41
  Day 8: H1N1 | 42.05 [27.89 to 63.40] | 185.61 [125.31 to 274.92] | 163.84 [101.76 to 263.81] | 319.86 [208.59 to 490.50]
  Day 181: H1N1: number analyzed (Participants) | 39 | 39 | 44 | 36
  Day 181: H1N1 | 67.55 [41.88 to 108.96] | 167.28 [121.35 to 230.59] | 74.14 [52.08 to 105.54] | 159.95 [104.34 to 245.20]
  Day 1 (Baseline): H3N2 | 53.68 [36.84 to 78.22] | 52.52 [37.35 to 73.85] | 50.59 [37.90 to 67.53] | 75.31 [50.06 to 113.30]
  Day 8: H3N2: number analyzed (Participants) | 41 | 42 | 44 | 41
  Day 8: H3N2 | 51.46 [37.34 to 70.91] | 211.76 [148.46 to 302.04] | 220.95 [155.08 to 314.81] | 345.29 [262.51 to 454.16]
  Day 181: H3N2: number analyzed (Participants) | 39 | 39 | 44 | 36
  Day 181: H3N2 | 67.50 [45.07 to 101.09] | 186.06 [136.00 to 254.55] | 158.74 [116.46 to 216.37] | 235.10 [167.17 to 330.64]
  Day 1 (Baseline): Victoria-lineage: number analyzed (Participants) | 41 | 43 | 44 | 40
  Day 1 (Baseline): Victoria-lineage | 113.97 [76.71 to 169.33] | 121.61 [86.46 to 171.06] | 91.41 [64.64 to 129.27] | 137.99 [95.73 to 198.91]
  Day 8: Victoria-lineage: number analyzed (Participants) | 41 | 42 | 44 | 41
  Day 8: Victoria-lineage | 34.65 [23.93 to 50.17] | 91.27 [68.41 to 121.78] | 113.14 [81.85 to 156.40] | 122.10 [88.63 to 168.20]
  Day 181: Victoria-lineage: number analyzed (Participants) | 39 | 39 | 44 | 36
  Day 181: Victoria-lineage | 37.59 [26.09 to 54.17] | 76.56 [55.37 to 105.87] | 72.27 [53.70 to 97.26] | 70.62 [48.32 to 103.19]
  Day 1 (Baseline): Yamagata-lineage | 113.13 [70.09 to 182.60] | 124.60 [86.34 to 179.83] | 84.47 [55.85 to 127.75] | 128.43 [81.44 to 202.53]
  Day 8: Yamagata-lineage: number analyzed (Participants) | 41 | 42 | 44 | 41
  Day 8: Yamagata-lineage | 54.68 [36.21 to 82.59] | 118.85 [90.96 to 155.29] | 116.79 [81.49 to 167.37] | 194.38 [141.31 to 267.38]
  Day 181: Yamagata-lineage: number analyzed (Participants) | 39 | 39 | 44 | 36
  Day 181: Yamagata-lineage | 55.08 [36.30 to 83.57] | 106.23 [79.98 to 141.08] | 69.87 [52.76 to 92.54] | 112.06 [73.69 to 170.39]

12. Secondary Outcome: Phase 1/2: GMFR of Anti-HA Antibodies at Days 8 and 181, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
  95% CI was calculated based on the difference in the log-transformed values for GMT, then back transformed to the original scale for presentation.
Time Frame: Day 1 (Baseline), Day 8 and Day 181
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug
Number analyzed (Participants) | 41 | 42 | 44 | 41
ratio
  Day 8: H1N1 | 0.78 [0.62 to 0.98] | 3.48 [2.35 to 5.14] | 4.30 [2.76 to 6.69] | 5.91 [3.83 to 9.11]
  Day 181: H1N1: number analyzed (Participants) | 39 | 39 | 44 | 36
  Day 181: H1N1 | 1.21 [0.87 to 1.67] | 2.99 [1.95 to 4.57] | 2.18 [1.51 to 3.14] | 2.92 [2.11 to 4.04]
  Day 8: H3N2 | 0.96 [0.73 to 1.25] | 4.21 [2.77 to 6.40] | 4.37 [2.73 to 6.99] | 4.58 [2.90 to 7.25]
  Day 181: H3N2: number analyzed (Participants) | 39 | 39 | 44 | 36
  Day 181: H3N2 | 1.27 [0.89 to 1.82] | 3.24 [2.37 to 4.41] | 3.27 [2.28 to 4.70] | 3.09 [2.14 to 4.46]
  Day 8: Victoria-lineage: number analyzed (Participants) | 41 | 42 | 44 | 40
  Day 8: Victoria-lineage | 0.30 [0.22 to 0.41] | 0.77 [0.54 to 1.10] | 1.24 [0.86 to 1.77] | 0.85 [0.55 to 1.30]
  Day 181: Victoria-lineage: number analyzed (Participants) | 39 | 39 | 44 | 35
  Day 181: Victoria-lineage | 0.34 [0.25 to 0.48] | 0.54 [0.37 to 0.80] | 0.82 [0.59 to 1.15] | 0.48 [0.32 to 0.70]
  Day 8: Yamagata-lineage | 0.48 [0.37 to 0.63] | 0.98 [0.72 to 1.32] | 1.38 [1.00 to 1.90] | 1.51 [1.05 to 2.17]
  Day 181: Yamagata-lineage: number analyzed (Participants) | 39 | 39 | 44 | 36
  Day 181: Yamagata-lineage | 0.53 [0.40 to 0.69] | 0.77 [0.56 to 1.07] | 0.96 [0.67 to 1.37] | 0.85 [0.66 to 1.09]

13. Secondary Outcome: Phase 2 NH and Phase 2 Extension: Percentage of Participants With Seroconversion, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B
Description: as for outcome 7
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 2 NH: mRNA-1010 12.5 ug: Participants received mRNA-1010 12.5 ug by IM injection on Day 1.
Arm/Group | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug | Phase 2 Extension: Afluria Quadrivalent 60 ug | Phase 2 Extension: mRNA-1010 6.25 ug | Phase 2 NH: mRNA-1010 12.5 ug | Phase 2 Extension: mRNA-1010 25 ug
Number analyzed (Participants) | 52 | 144 | 138 | 141 | 48 | 49 | 47 | 46
Percentage of participants
  H1N1 | 59.6 [45.10 to 72.99] | 72.2 [64.15 to 79.36] | 84.8 [77.68 to 90.33] | 85.8 [78.95 to 91.12] | 50.0 [35.23 to 64.77] | 59.2 [44.21 to 73.00] | 68.1 [52.88 to 80.91] | 73.9 [58.87 to 85.73]
  H3N2 | 40.4 [27.01 to 54.90] | 66.0 [57.62 to 73.65] | 71.7 [63.45 to 79.07] | 78.7 [71.04 to 85.16] | 43.8 [29.48 to 58.82] | 44.9 [30.67 to 59.77] | 66.0 [50.69 to 79.14] | 80.4 [66.09 to 90.64]
  Victoria-lineage | 32.7 [20.33 to 47.11] | 22.9 [16.33 to 30.65] | 33.3 [25.54 to 41.86] | 37.1 [29.13 to 45.71] | 47.9 [33.29 to 62.81] | 10.2 [3.40 to 22.23] | 21.7 [10.95 to 36.36] | 28.3 [15.99 to 43.46]
  Yamagata-lineage | 32.7 [20.33 to 47.11] | 41.7 [33.52 to 50.17] | 47.8 [39.26 to 56.49] | 51.8 [43.21 to 60.26] | 47.9 [33.29 to 62.81] | 24.5 [13.34 to 38.87] | 43.5 [28.93 to 58.89] | 39.1 [25.09 to 54.63]

14. Secondary Outcome: Phase 2 NH and Phase 2 Extension: GMFR of Anti-HA Antibodies at Day 29, as Measured by HAI Assay for Vaccine-Matched Seasonal Influenza A and B Strains
Description: as for outcome 8
Time Frame: Day 29
Population: PP Set: consisted of all participants who received the investigational product and who complied with the injection schedule and timing of immunogenicity blood sampling, did not have influenza infection at baseline through Day 29, and had no major protocol deviations that impacted the immune response. Number Analyzed = participants who were evaluable at specified timepoints. Number Analyzed = participants who were evaluable at specified timepoints.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug | Phase 2 Extension: Afluria Quadrivalent 60 ug | Phase 2 Extension: mRNA-1010 6.25 ug | Phase 2 Extension: mRNA-1010 12.5 ug | Phase 2 Extension: mRNA-1010 25 ug
Number analyzed (Participants) | 52 | 144 | 138 | 141 | 48 | 49 | 47 | 46
ratio
  H1N1 | 4.19 [2.82 to 6.23] | 7.64 [6.22 to 9.38] | 12.15 [9.38 to 15.73] | 11.96 [9.81 to 14.58] | 6.08 [3.84 to 9.64] | 6.03 [4.22 to 8.61] | 7.21 [4.90 to 10.63] | 12.58 [7.95 to 19.90]
  H3N2 | 3.17 [2.20 to 4.58] | 6.28 [5.02 to 7.84] | 8.17 [6.63 to 10.06] | 8.70 [7.22 to 10.48] | 3.78 [2.56 to 5.58] | 4.51 [3.15 to 6.46] | 6.66 [4.57 to 9.69] | 9.30 [6.11 to 14.17]
  Victoria-lineage: number analyzed (Participants) | 52 | 144 | 138 | 141 | 48 | 49 | 46 | 46
  Victoria-lineage | 3.30 [2.13 to 5.11] | 2.27 [2.00 to 2.58] | 3.06 [2.60 to 3.60] | 2.79 [2.47 to 3.15] | 3.91 [2.66 to 5.76] | 1.69 [1.30 to 2.20] | 1.84 [1.39 to 2.43] | 2.47 [1.76 to 3.46]
  Yamagata-lineage: number analyzed (Participants) | 52 | 144 | 138 | 141 | 48 | 49 | 46 | 46
  Yamagata-lineage | 3.07 [2.19 to 4.29] | 3.33 [2.85 to 3.90] | 3.73 [3.09 to 4.51] | 3.67 [3.15 to 4.27] | 3.72 [2.70 to 5.15] | 2.29 [1.67 to 3.14] | 3.03 [2.18 to 4.21] | 3.08 [2.08 to 4.55]

15. Secondary Outcome: Phase 2 NH and Phase 2 Extension: Percentage of Participants With HAI Titer ≥1:40 at Day 29
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug | Phase 2 Extension: Afluria Quadrivalent 60 ug | Phase 2 Extension: mRNA-1010 6.25 ug | Phase 2 Extension: mRNA-1010 12.5 ug | Phase 2 Extension: mRNA-1010 25 ug
Number analyzed (Participants) | 52 | 144 | 138 | 141 | 48 | 49 | 47 | 46
percentage of participants
  H1N1 | 92.3 [81.46 to 97.86] | 97.2 [93.04 to 99.24] | 97.1 [92.74 to 99.20] | 98.6 [94.97 to 99.83] | 95.8 [85.75 to 99.49] | 93.9 [83.13 to 98.72] | 95.7 [85.46 to 99.48] | 97.8 [88.47 to 99.94]
  H3N2 | 90.4 [78.97 to 96.80] | 91.0 [85.06 to 95.11] | 91.3 [85.30 to 95.43] | 91.5 [85.61 to 95.52] | 81.3 [67.37 to 91.05] | 89.8 [77.77 to 96.60] | 93.6 [82.46 to 98.66] | 97.8 [88.47 to 99.94]
  Victoria-lineage: number analyzed (Participants) | 52 | 141 | 138 | 141 | 48 | 49 | 47 | 46
  Victoria-lineage | 96.2 [86.79 to 99.53] | 91.7 [85.90 to 95.62] | 90.6 [84.43 to 94.89] | 91.4 [85.51 to 95.49] | 100.0 [92.60 to 100.0] | 75.5 [61.13 to 86.66] | 89.1 [76.43 to 96.38] | 82.6 [68.58 to 92.18]
  Yamagata-lineage | 96.2 [86.79 to 99.51] | 99.3 [96.19 to 99.98] | 96.4 [91.75 to 98.81] | 97.2 [92.90 to 99.22] | 97.9 [88.93 to 99.95] | 93.9 [83.13 to 98.72] | 95.7 [85.16 to 99.47] | 91.3 [79.21 to 97.58]

ADVERSE EVENTS:
Time Frame: Up to 6 months (Day 181, end of study)
Description: Safety Analysis Set consisted of all randomly assigned participants who received the investigational product. Participants were included in the vaccination group corresponding to the study injection they actually received.
  Note, not all solicited ARs were considered AEs. The Investigator reviewed whether the solicited AR was also to be recorded as an AE.
Arm/Group | Phase 1/2: Placebo | Phase 1/2: mRNA-1010 50 ug | Phase 1/2: mRNA-1010 100 ug | Phase 1/2: mRNA-1010 200 ug | Phase 2 NH: Afluria Quadrivalent 60 ug | Phase 2 NH: mRNA-1010 25 ug | Phase 2 NH: mRNA-1010 50 ug | Phase 2 NH: mRNA-1010 100 ug | Phase 2 Extension: Afluria Quadrivalent 60 ug | Phase 2 Extension: mRNA-1010 6.25 ug | Phase 2 Extension: mRNA-1010 12.5 ug | Phase 2 Extension: mRNA-1010 25 ug
All-Cause Mortality (participants affected / at risk) | 1/45 | 0/45 | 0/46 | 0/44 | 0/54 | 0/150 | 0/147 | 1/147 | 0/51 | 1/50 | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/45 | 0/45 | 0/46 | 1/44 | 1/54 | 3/150 | 5/147 | 4/147 | 1/51 | 2/50 | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 26/45 | 39/45 | 44/46 | 42/44 | 37/54 | 130/150 | 133/147 | 133/147 | 33/51 | 45/50 | 38/50 | 45/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1/2: Placebo (N=45) | Phase 1/2: mRNA-1010 50 ug (N=45) | Phase 1/2: mRNA-1010 100 ug (N=46) | Phase 1/2: mRNA-1010 200 ug (N=44) | Phase 2 NH: Afluria Quadrivalent 60 ug (N=54) | Phase 2 NH: mRNA-1010 25 ug (N=150) | Phase 2 NH: mRNA-1010 50 ug (N=147) | Phase 2 NH: mRNA-1010 100 ug (N=147) | Phase 2 Extension: Afluria Quadrivalent 60 ug (N=51) | Phase 2 Extension: mRNA-1010 6.25 ug (N=50) | Phase 2 Extension: mRNA-1010 12.5 ug (N=50) | Phase 2 Extension: mRNA-1010 25 ug (N=49)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic amnestic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Distributive shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1/2: Placebo (N=45) | Phase 1/2: mRNA-1010 50 ug (N=45) | Phase 1/2: mRNA-1010 100 ug (N=46) | Phase 1/2: mRNA-1010 200 ug (N=44) | Phase 2 NH: Afluria Quadrivalent 60 ug (N=54) | Phase 2 NH: mRNA-1010 25 ug (N=150) | Phase 2 NH: mRNA-1010 50 ug (N=147) | Phase 2 NH: mRNA-1010 100 ug (N=147) | Phase 2 Extension: Afluria Quadrivalent 60 ug (N=51) | Phase 2 Extension: mRNA-1010 6.25 ug (N=50) | Phase 2 Extension: mRNA-1010 12.5 ug (N=50) | Phase 2 Extension: mRNA-1010 25 ug (N=49)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epiretinal membrane (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 3 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 8 | 18 | 17 | 5 | 23 | 31 | 30 | 3 | 4 | 6 | 11
Chills (General disorders) | 2 | 14 | 26 | 31 | 6 | 44 | 52 | 73 | 8 | 9 | 5 | 18
Fatigue (General disorders) | 10 | 24 | 40 | 35 | 16 | 79 | 86 | 96 | 16 | 23 | 20 | 27
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 1 | 6 | 4 | 4 | 2 | 0 | 0 | 1
Injection site dermatitis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 2 | 6 | 1 | 1 | 8 | 5 | 11 | 0 | 1 | 3 | 0
Injection site induration (General disorders) | 0 | 3 | 4 | 1 | 1 | 9 | 12 | 14 | 1 | 0 | 4 | 2
Injection site lymphadenopathy (General disorders) | 3 | 11 | 16 | 22 | 10 | 40 | 45 | 52 | 7 | 13 | 14 | 16
Injection site pain (General disorders) | 7 | 33 | 40 | 40 | 17 | 110 | 120 | 122 | 25 | 37 | 32 | 41
Pyrexia (General disorders) | 0 | 2 | 11 | 13 | 2 | 10 | 14 | 25 | 0 | 0 | 2 | 3
Seasonal allergy (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 2 | 3 | 8 | 17 | 19 | 21 | 1 | 5 | 3 | 3
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 0 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3 | 3 | 4 | 0 | 2 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 2 | 1 | 5 | 8 | 8 | 8 | 0 | 3 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 10 | 28 | 27 | 11 | 57 | 68 | 73 | 10 | 12 | 13 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 18 | 36 | 31 | 12 | 72 | 88 | 98 | 14 | 16 | 16 | 28
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 19 | 29 | 33 | 10 | 78 | 79 | 82 | 20 | 21 | 18 | 24
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 3 | 7 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 5 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 5 | 4 | 7 | 1 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 4 | 0 | 0 | 3 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 4 | 0 | 1 | 3 | 2
Subgaleal haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04956575/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04956575/SAP_001.pdf